CLINICAL TRIAL: NCT03362931
Title: A Prospective, Multicenter Clinical Trial Designed to Evaluate the Safety and Effectiveness of the XEN45 Glaucoma Treatment System in Patients With Angle Closure Glaucoma
Brief Title: Safety and Effectiveness of the XEN45 Glaucoma Treatment System in Patients With Angle Closure Glaucoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1924-701-007
Record Dates: First submitted 2017-11-30; First posted 2017-12-05 (Actual); Results first posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-04

CONDITIONS: Glaucoma; Angle-Closure
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- XEN45 Glaucoma Treatment System (hereafter referred to as XEN) (Experimental): XEN45 unilaterally implanted in the study eye
  Interventions: Device: XEN45

INTERVENTIONS:
Device: XEN45 — XEN45 unilaterally implanted in the study eye

SUMMARY:
This study will evaluate the safety and IOP-lowering effectiveness of XEN in patients with Angle Closure Glaucoma.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria: - Diagnosis of ACG defined as areas of iridotrabecular contact present in ≥ 2 quadrants and glaucomatous damage to optic disc and visual field, in the study eye - Study eye has healthy, free, and mobile conjunctiva in the target quadrant Exclusion Criteria: - Uncontrolled systemic disease (eg, diabetes, hypertension) - Known history of bleeding disorder or prolonged bleeding after surgery or those on pharmacologic blood thinners other than aspirin (up to 100 mg/day) - History of dermatologic keloid formation - Open angle glaucoma, active acute angle closure attack, congenital glaucoma, juvenile glaucoma, secondary glaucoma in the study eye - History of following surgeries in the study eye: o incisional refractive surgery (eg, radial keratotomy), other than astigmatic keratotomy or limbal relaxing incisions o corneal graft including partial grafts such as Descemet's stripping endothelial keratoplasty and Descemet's membrane endothelial keratoplasty o previous laser or incisional intraocular surgery that might interfere with the outcome of this trial - Previous glaucoma shunt implantation in the target quadrant in the study eye - Active or history of chronic uveitis in the study eye - Unable to discontinue contact lens wear in the study eye during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2022-03-18 (Actual); Study Completion 2022-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ALLERGAN INC., Study Director — Allergan
Locations (16):
- Australia (3):
  - Marsden Eye Specialists Parramatta /ID# 232761, Paramatta, New South Wales
  - Melbourne Eye Specialists /ID# 232767, Fitzroy, Victoria
  - Eye Surgery Associates P/L ATF Eye Surgery Associates Unit Trust /ID# 232765, Vermont South, Victoria
- Canada (3):
  - Institut de loeil des Laurentides /ID# 232780, Boisbriand, Quebec
  - Ophthalmology Clinic Bellevue /ID# 232782, Montreal, Quebec
  - Prism Eye Institute /ID# 232917, Mississauga
- Singapore (2):
  - Nuh Medical Centre /ID# 232905, Singapore
  - Tan Tock Seng Hospital /ID# 233014, Singapore
- Seoul National University Hospital /ID# 233099, Seoul, South Korea
- Taiwan (2):
  - Buddhist Tzu Chi General Hospital /ID# 232664, Hualien City, Hualien
  - Taipei Veterans General Hospital /ID# 232948, Taipei City, Taipei
- United Kingdom (5):
  - Royal Surrey County Hospital /ID# 233028, Guildford, England
  - Manchester University NHS Foundation Trust /ID# 232808, Manchester, Lancashire
  - Queen Victoria Hospital /ID# 232812, East Grinstead, West Sussex
  - East Suffolk and North Essex NHS Foundation Trust /ID# 232804, Colchester
  - NHS Lothian /ID# 233052, Edinburgh

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing, please refer to the link below
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: XEN45 Glaucoma Treatment System (Hereafter Referred to as XEN): XEN45 unilaterally implanted in the study eye
Period: Overall Study
Arm/Group | Experimental: XEN45 Glaucoma Treatment System (Hereafter Referred to as XEN)
Started | 62
Completed | 59
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | XEN45 Glaucoma Treatment System (Hereafter Referred to as XEN)
Number analyzed (Participants) | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.0 (9.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 62
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 31
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 8
  South Korea | 3
  Singapore | 10
  Taiwan | 9
  United Kingdom | 7
  Australia | 25

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving at Least a 20% Reduction From Baseline Hour 0 IOP While on the Same Number or Fewer IOP Lowering Medications at Month 12
Description: IOP will be measured using a Goldmann applanation tonometer
Time Frame: Month 12
Population: Implanted population, defined as all subjects implanted with XEN45, with data at visit. (Missing data and data after the 1st non-study surgical procedures for IOP control or device explant are not counted or imputed.)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | XEN45 Glaucoma Treatment System (Hereafter Referred to as XEN)
Number analyzed (Participants) | 56
percentage of participants | 80.5 [68.4 to 88.8]

2. Secondary Outcome: Change From Baseline the Number of Concomitant IOP-lowering Medications
Description: The number of concomitant IOP-lowering medications following implantation will be compared with the number prior to implantation.
Time Frame: Month 12
Population: Implanted population, defined as all subjects implanted with XEN45, with data at visit.
Measure: Mean (Standard Deviation); unit: Number of medications in study eye
Arm/Group | XEN45 Glaucoma Treatment System (Hereafter Referred to as XEN)
Number analyzed (Participants) | 56
Number of medications in study eye | -1.6 (1.33)

ADVERSE EVENTS:
Time Frame: Up tp 12 months after the initiation of XEN45 Implant related procedures
Arm/Group | Experimental: XEN45 Glaucoma Treatment System (Hereafter Referred to as XEN)
All-Cause Mortality (participants affected / at risk) | 2/62
Serious Adverse Events (participants affected / at risk) | 12/62
Other Adverse Events (participants affected / at risk) | 44/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: XEN45 Glaucoma Treatment System (Hereafter Referred to as XEN) (N=62)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 (1)
ANGLE CLOSURE GLAUCOMA (Eye disorders) | 1 (1)
CONJUNCTIVAL EROSION (Eye disorders) | 3 (3)
SUBCONJUNCTIVAL FIBROSIS (Eye disorders) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1)
SEPTIC SHOCK (Infections and infestations) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (1)
SKIN LACERATION (Injury, poisoning and procedural complications) | 1 (1)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1)
INTRAOCULAR PRESSURE INCREASED (Investigations) | 1 (1)
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1)
DEVICE PHYSICAL PROPERTY ISSUE (Product Issues) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1)
CALCULUS BLADDER (Renal and urinary disorders) | 1 (1)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HYPOTENSION (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: XEN45 Glaucoma Treatment System (Hereafter Referred to as XEN) (N=62)
CHOROIDAL EFFUSION (Eye disorders) | 5 (5)
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 6 (6)
CONJUNCTIVAL HYPERAEMIA (Eye disorders) | 13 (18)
CONJUNCTIVAL OEDEMA (Eye disorders) | 6 (8)
CORNEAL OEDEMA (Eye disorders) | 4 (5)
DRY EYE (Eye disorders) | 5 (6)
ERYTHEMA OF EYELID (Eye disorders) | 4 (6)
EYE PAIN (Eye disorders) | 4 (5)
EYELID OEDEMA (Eye disorders) | 4 (5)
FOREIGN BODY SENSATION IN EYES (Eye disorders) | 4 (4)
PUNCTATE KERATITIS (Eye disorders) | 5 (7)
VISION BLURRED (Eye disorders) | 4 (4)
VISUAL ACUITY REDUCED (Eye disorders) | 6 (6)
HYPHAEMA (Injury, poisoning and procedural complications) | 4 (4)
INTRAOCULAR PRESSURE INCREASED (Investigations) | 25 (33)
DEVICE OCCLUSION (Product Issues) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2017-10-04): https://cdn.clinicaltrials.gov/large-docs/31/NCT03362931/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-14): https://cdn.clinicaltrials.gov/large-docs/31/NCT03362931/SAP_001.pdf